CLINICAL TRIAL: NCT04746625
Title: Safety and Performance of the Polaris® 24 Adjustable Valve System in Hydrocephalus Patients' Treatment
Acronym: SAPPHYRE
Status: Recruiting | Type: Observational
Sponsor: Sophysa (Industry)
Responsible Party: Sponsor
Other Study IDs: PCLI 470-01
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; Adjustable valve; Polaris 24; Cerebrospinal fluid
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SAPPHYRE study is an ambispective (retrospective and prospective) PMCF study with the objective to evaluate the safety and performance of the Polaris® 24 adjustable valve system in the treatment of 126 patients with hydrocephalus.

DETAILED DESCRIPTION:
The SAPPHYRE study is an ambispective (retrospective and prospective), non-interventional, multicenter, post-market clinical follow-up study. The study objective is to evaluate the safety and performance of Sophysa's CE marked Polaris® 24 adjustable valve system in the treatment of hydrocephalus by shunting the cerebrospinal fluid. It is expected to recruit 126 patients in two-year. Patients will be followed-up up to 5 years post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with the Polaris® 24 adjustable valve system for the following reasons:

  * Primo implant of a valve shunt-based derivation system, or as a
  * Replacement of another valve -based shunt system, or
  * Endoscopic ventriculostomy (EVT) failure
* Patient having given his/her informed consent prior to inclusion in this study, as per local regulations

Exclusion Criteria:

* Confirmed or suspected infections along the length of the shunt (meningitis, ventriculitis, peritonitis, septicemia or bacteremia) or any infection present in any part of the body
* Patient on anticoagulant therapy, or presenting with bleeding diathesis, or with haemorrhagic CSF, as the presence of blood in the system could lead to an obstruction in the system
* Ventriculo-atrial shunts in patient suffering from congenital cardiopathies or other malformations of the cardio-pulmonary system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults, children and neonates, regardless of gender with hydrocephalus.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Device-related SAE / complications | 1 year
  Primary safety outcome will be assessed by the incidence of device-related serious adverse events / complications
Valve replacement | 1 year
  Primary performance outcome will be assessed by the incidence of valve replacements

SECONDARY OUTCOMES:
All adverse events / complications | Two (2) years post procedure, and yearly thereafter, up to five (5) years post implantation
  Long term safety will be assessed by the incidence of all adverse events/complications
Valve replacement | Two (2) years post procedure, and yearly thereafter, up to five (5) years post implantation
  Incidence of valve replacements
Implant procedure success | 0 day (post-procedure)
  Implant procedure success, defined as no immediate re-intervention post-procedure
Change of clinical status scores | One (1) year, two (2) years, and yearly thereafter, up to five (5) years post implantation
  Improvement of the following clinical status scores compared to baseline: the Modified Rankin Scale (for adults and children) and the Lansky Performance Scale (for children < 16 years old only)
Evolution of Clinical symptoms | One (1) year, two (2) years, and and yearly thereafter, up to five (5) years post implantation
  Clinical symptoms will be assessed according to a 4-grade scale (excellent, good, unchanged, worsened)
MRI stability | One (1) year, two (2) years, and yearly thereafter, up to five (5) years post implantation
  MRI (1.5Tesla or 3Tesla) stability of the pressure adjustment
Valve pressure adjustment | (if applicable), throughout the follow-up period: One (1) year, two (2) years, and and yearly thereafter, up to five (5) years post implantation
  If required by patient's condition, the physician will adjust the valve pressure with the adjustment kit provided with the Polaris 24 valve. Physician will evaluate the ease of reading and adjusting of the valve pressure (from easy to difficult)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Scavarda, Prof, Principal Investigator — La Timone Children's Hospital - Paediatrics Neurosurgery Department
Locations (2):
- France (2):
  - La Timone Children's Hospital, Marseille
  - La Pitié Salpétrière Hospital, Paris

REFERENCES:
- See also: Sponsor's website — http://www.sophysa.com